CLINICAL TRIAL: NCT00963742
Title: Lenstec Softec HD Posterior Chamber Intraocular Lens (PCIOL) Clinical Investigational Protocol
Brief Title: Lenstec Softec HD Posterior Chamber Intraocular Lens Clinical Investigational Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE G060058
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cataract
Keywords: cataract surgery; IOL; Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenstec Softec HD IOL implantation (Experimental): 390 eyes of 390 study subjects all receiving the investigational IOL; IOL implanted after surgical removal of cataract
  Interventions: Device: Lenstec Softec HD IOL implantation

INTERVENTIONS:
Device: Lenstec Softec HD IOL implantation — surgical removal of cataract and implantation of Softec HD PCIOL
  Other Names: Softec HD PCIOL; Softec HD Posterior Chamber IOL; Softec HD Posterior Chamber Intraocular Lens

SUMMARY:
The objectives of this multi-center clinical investigation are to determine the safety and effectiveness of the Lenstec Softec HD Posterior Chamber intraocular lens (IOL) following one year of post-operative assessment.

DETAILED DESCRIPTION:
The Softec HD Posterior Chamber IOL is designed for the treatment of aphakia. The lens is indicated for primary implantation when a cataractous lens has been removed by phacoemulsification with circular tear capsulotomy and the posterior capsule intact. The intended benefit of the Softec HD Posterior Chamber IOL is to provide enhanced vision.

ELIGIBILITY:
Inclusion Criteria:

* Cataract requiring cataract extraction
* Study IOL to only be implanted in 1 eye
* Distance BCVA 20/40 or worse or glare acuity worse than 20/30
* Ability to comply with study follow-up requirements

Exclusion Criteria:

* Patients with serious corneal disease, previous surgery or serious systemic disease
* Ocular condition that could impact vision after cataract surgery
* Pregnant or lactating women
* Use of ocular or systemic medications that could impact vision

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Distance Best Corrected Visual Acuity | 1 year

SECONDARY OUTCOMES:
FDA IOL Grid Adverse Events | through 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sanders, M.D. Ph.D, Study Director — Center for Clinical Research